CLINICAL TRIAL: NCT06094010
Title: A Phase IIIb Multicenter, Single-Arm, Open-Label Surveillance Study of Susceptibility to Baloxavir Marboxil in Pediatric Patients With Influenza and Transmission of Influenza to Household Contacts
Brief Title: A Surveillance Study of Susceptibility to Baloxavir Marboxil in Pediatric Participants With Influenza and Transmission of Influenza to Household Contacts
Acronym: Pebblestone
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV44536; 2023-504672-22-00 (EU CTIS Number)
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — baloxavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Baloxavir Marboxil (Experimental): Participants will receive a single oral dose of baloxavir marboxil on Day 1 (based on body weight and age). HHCs related to IPs will be enrolled but will not receive treatment.
  Interventions: Drug: Baloxavir Marboxil

INTERVENTIONS:
Drug: Baloxavir Marboxil — Baloxavir marboxil will be administered as an oral suspension per body weight (≥80 kilograms (kg): 80 milligrams (mg); ≥20 kg to < 80 kg: 40 mg; <20 kg: 2 mg/kg).

SUMMARY:
This study consists of two parts: Part A Surveillance and Part B Transmission.

The main purpose of Part A is to evaluate the prevalence of pre-dose and treatment-emergent amino acid substitutions in pediatric participants' susceptibility <12 years with influenza treated with baloxavir marboxil.

Part B will include a subset of Part A participants who have household contacts (HHCs) recruited to the study. Part B will evaluate the incidence of onward influenza transmission from pediatric index participants (IPs) under 5 years of age and those aged 5 to under 12 years, treated with baloxavir marboxil, to their HHCs.

ELIGIBILITY:
Inclusion Criteria (Part A):

* Participants with symptoms suggestive of influenza based on investigator's judgement with diagnosis confirmed by a positive local influenza test within 24 hours before full study screening
* Participants with a negative severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test within 48 hours before full study screening
* Time interval between onset of influenza symptoms and the pre-dose examinations at screening is 48 hours or less

Inclusion Criteria (Part B):

[A] IP:

* Eligible to take part in Part A
* Lives in a household with a HHC willing to be recruited as full household contact

[B] HHCs:

- Each HHC living in the home of an IP at the time of IP treatment must be screened for partial or full-study HHC eligibility

[C] Partial HHC:

* Starts screening within 1 calendar day after IP treatment
* Negative influenza and SARS-CoV-2 test at screening after IP's treatment with baloxavir marboxil
* HHC lives in a household where 1 or more HHCs meet the full-study HHC requirements AND at least 1 full-study HHC has not received the influenza vaccine within 6 months prior to screening
* HHC lives in a household where 1 or more HHCs meet the full-study HHC requirements AND at least 1 full-study HHC has not received the influenza vaccine within 6 months prior to screening.
* HHC lives with other HHCs (if applicable) who fulfill all the "Partial household contact" criteria

[D] Full-study HHC:

* Fulfills the "Partial household contact" criteria
* Agrees to participate in the full study
* Will reside in the IP's house for at least 12 of the next 15 days and will be present for scheduled study visits
* No influenza symptoms within 7 days prior to screening
* Does not have a moderate or worse active infections OR infections requiring systemic or otherwise internally administered or otherwise internally administered antibiotic/antiviral/antifungal therapy

Exclusion Criteria (Part A):

* Participants with severe influenza virus infection requiring inpatient treatment
* Severely immunocompromised participants [including participants receiving immunosuppressant therapy, or those with cancer or human immunodeficiency virus (HIV) infection] as defined by the investigator
* Participants with concurrent (non-influenza) infections requiring systemic anti-microbial and/or anti-viral therapy at the pre-dose examinations
* Treatment with baloxavir marboxil, peramivir, laninamivir, oseltamivir, zanamivir, rimantadine, umifenovir or amantadine within 30 days prior to screening
* Treatment with an investigational influenza-specific monoclonal antibody within 6 months or 5 half-lives, whichever is longer, prior to screening
* Treatment with an investigational therapy within 30 days or 5 half-lives, whichever is longer, prior to screening
* Known hypersensitivity to baloxavir marboxil or the drug product excipients
* Females who have commenced menarche (i.e., child-bearing potential)

Exclusion Criteria (Part B):

* IPs who fulfill an exclusion criterion for Part A
* HHCs deemed to require influenza post-exposure prophylaxis with influenza antiviral treatment due to their risk of developing influenza-related complications in accordance with local guidelines or clinical practice
* HHCs diagnosed with influenza by health care professional in the past 4 weeks

Ages: 3 Weeks to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 750 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2027-05-11 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Part A: Percentage of Participants With Resistance-associated Pre-treatment Substitutions | Day 1 (Baseline)
Part A: Percentage of Participants With Resistance-associated Treatment-emergent Substitutions | Days 4, 6 and 10

SECONDARY OUTCOMES:
Part A: Percentage of IPs With Resistance-associated Treatment-emergent Substitutions by Age Groups (<5 Years [< 1 Year, ≥ 1 Year to < 5 Years], and 5 to < 12 Years) | Days 4, 6 and 10
Part A: Percentage of IPs With Novel Treatment-emergent Mutations in Polymerase Acidic Protein (PA) | Days 4, 6 and 10
Part A: Percentage of IPs With Resistance-associated Treatment-emergent Substitutions by Baseline Vaccination Status | Days 4, 6 and 10
Part A: Percentage of IPs With Influenza Virus Type (A or B) and Subtype (A/H1 or A/H3) | Day 1 (Baseline)
Part A: Change From Baseline in Viral Titers by Quantitative Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) | Baseline (Day 1); Days 4, 6 and 10
Part A: Susceptibility to Baloxavir Marboxil by Phenotyping of Virus With Novel Genotypic PA Substitutions | Days 4, 6 and 10
Part A: Number of IPs with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 29
  AEs were reported according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0).
Part B: Percentage of HHCs With Transmission of Influenza Virus by Confirmed by Central RT-PCR, With Virus Subtype Consistent With the IP | Day 6, Day 10
Part B: Percentage of HHCs Who Develops Influenza Symptoms With Transmission of Influenza Virus Confirmed by Central RT-PCR, With Virus Subtype Consistent With the IP | Day 6, Day 10

OTHER OUTCOMES:
Percentage of HHCs Who Become PCR (+) for Influenza Bearing a PA/I38X Substitution (or Other Identified Substitution) Including All Data up to Day 15 | Up to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (51):
- United States (28):
  - Central Alabama Research, Birmingham, Alabama
  - Harrisburg Family Medical Center, Harrisburg, Arkansas
  - Kendall South Medical Center Inc., Miami, Florida
  - Avanza Medical Research Center, Pensacola, Florida
  - Tekton Research - Chamblee Georgia, Chamblee, Georgia
  - Tekton Research Lawrenceville, Lawrenceville, Georgia
  - Velocity Clinical Research at Primary Pediatrics Macon, Macon, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Mishawaka Osteopathic Clinic, Mishawaka, Indiana
  - Kentucky Pediatric Research Center, Bardstown, Kentucky
  - Velocity Clinical Research Lafayette, Lafayette, Louisiana
  - Velocity Clinical Research, Slidell, Slidell, Louisiana
  - Velocity Clinical Research, Grand Island, Grand Island, Nebraska
  - Machuca Family Medicine, Las Vegas, Nevada
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Helios Clinical Research, Inc (former Ventavia Research Group), Middleburg Heights, Ohio
  - Frontier Clinical Research, Smithfield, Pennsylvania
  - Coastal Pediatric Research, Charleston, South Carolina
  - Tekton Research - Beaumont, Beaumont, Texas
  - Oak Cliff Research Company, LLC, Dallas, Texas
  - Mercury Clinical Research, Houston, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Oak Cliff Research Company, LLC, Richardson, Texas
  - Sun Research Institute, San Antonio, Texas
  - Tekton Research, San Antonio, Texas
  - Siena Research Network, Sugar Land, Texas
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Frontier Clinical Research, LLC, Kingwood, West Virginia
- Bulgaria (8):
  - Medical Centre "Asklepii", OOD, Dupnitsa
  - MHAT " St. Ivan Rilski " Kozloduy, Kozloduy
  - MHAT Stamen Iliev AD, Montana
  - MHAT City Clinic - Saint George, Montana
  - SHATPPD Dr. Dimitar Gramatikov, Ruse Ltd., Rousse
  - MHAT Sliven - Military Medial Academy, Sliven
  - AGPSMP Pediatric diseases South park OOD, Sofia
  - Medical Center Hera Sofia, Sofia
- Poland (11):
  - NZOZ Salmed, ??czna
  - Centrum Medyczne K2J2, ?ód?
  - IN VIVO Sp. z o.o., Bydgoszcz
  - NZOZ Vitamed, Bydgoszcz
  - Centrum Medyczne Pratia Cz?stochowa, Cz?stochowa
  - Niepubliczny Zaklad Opieki Zdrowotnej "Amed", Grójec
  - Vita Longa Sp. z o.o., Katowice
  - NZLA Michalkowice Rybarczyk i partnerzy, Spolka Lekarska, Siemianowice ?l?skie
  - Jaroslaw Kierkus Prywatna Prakyka Lekarska, Warsaw
  - Centrum Medyczne K2J2, Wo?omin
  - Vistamed & Vertigo Spó?Ka Z Ograniczon? Odpowiedzialno?Ci?, Wroc?aw
- Spain (4):
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, LA Coruna
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing